CLINICAL TRIAL: NCT02717364
Title: Yervoy® Postmarketing Surveillance for Patients in Japan With Unresectable, Malignant Melanoma
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA184-438
Record Dates: First submitted 2016-02-16; First posted 2016-03-23 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Population With Yervoy Exposure: Population With Yervoy Exposure

SUMMARY:
This study is a local, prospective, non-interventional, non-controlled, multicenter, observational study (regulatory postmarketing surveillance). Each physician will enroll patients who have received at least 1 dose of Yervoy, and each patient will be followed for up to 12 months. All patients will be evaluated for safety and effectiveness during Yervoy use (4 doses) and for 12 months from the first dose of Yervoy to confirm the safety profile of Yervoy under routine, daily practice

ELIGIBILITY:
Inclusion Criteria:

* All patients who are initiating treatment with Yervoy

Exclusion Criteria:

* Not Applicable

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) by types among the analysis population | 12 months
The Overall Survival (OS) Rate | 12 months
The factors that potentially affect safety or effectiveness | 12 months
  Stratified analysis on the incidence of adverse events (AEs) and effectiveness by patient background

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Chiyoda-ku, Tokyo
  - Local Institution, Tokyo

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome